# **Informed Consent Form**

Alcohol Health Education With Personalized Feedback Boosters

NCT03440463

Last updated: 1/19/2018

# INFORMED CONSENT DOCUMENT OLD DOMINION UNIVERSITY

PROJECT TITLE: Alcohol Health Education with Personalized Feedback Boosters 2

## INTRODUCTION

The purposes of this form are to give you information that may affect your decision whether to say YES or NO to participation in this research and to record the consent of those who say YES. Project Alcohol Health Education with Personalized Feedback Boosters assesses alcohol health behaviors and related constructs over an extended period of time. The project takes place in room 234 in the Mills Godwin Building.

#### **RESEARCHERS**

Abby L. Braitman, Ph.D., Research Associate, Psychology, College of Sciences, Responsible Project Investigator, <a href="mailto:abraitma@odu.edu">abraitma@odu.edu</a>, 132-B Mills Godwin Building

Michelle L. Kelley, Ph.D., Professor, Chair, Psychology, College of Sciences, Co-Investigator, <a href="mailto:mkelley@odu.edu">mkelley@odu.edu</a>, 134-C Mills-Godwin Building, 757-683-4459

#### **DESCRIPTION OF RESEARCH STUDY**

Several studies have been conducted looking into the subject of student health behaviors related to drinking. The current study investigates the effects of a brief computerized education session on student drinking behaviors over an extended period of time.

If you decide to participate, then you will join a study involving assessment of your own health behaviors. If you say YES, then you will complete a computerized survey (approximately 45 to 60 minutes) assessing your current health behaviors. This would be followed by approximately 30-45 minutes of exposure to a computerized intervention and would take place room 234 in the Mills Godwin Building. After completing this first appointment, you may be eligible for additional assessments for monetary compensation. If you complete this baseline procedure plus both follow-up assessments, your total participation time for the project will be approximately 2 hours and 30 minutes to 3 hours (depending on how long it takes you to complete each survey). Approximately 600 ODU students will be participating in this study.

#### **EXCLUSIONARY CRITERIA**

within the past 14 days, you are not eligible for this study.

You must be between at least 18 years old but not older than 24 years old to be eligible for this study. In addition, you must have consumed at least 1 alcoholic drink within the past 2 weeks. If you have not consumed alcohol

# **RISKS AND BENEFITS**

RISKS: If you decide to participate in this study, it is possible you may experience some discomfort answering questions regarding your behaviors and actions. If you would like to speak to someone at Counseling Services you may call 757-683-4401 or go to 1526 Webb Center. The research involves using a computer, so the risks involved with that are similar to typical computer use.

Additionally, identifying information will be collected from each participant. Alcohol use is illegal for individuals under 21, and so all efforts will be made to safeguard your information. Files with identifying information will be kept only on an encrypted external storage device, and that device will be kept in locked storage location when not in use. Hardcopies of signed informed consent documents will be kept in a locked filing cabinet. If you are using public computers owned and operated by ODU there may be the possibility of institutional monitoring of your responses. And, as with any research, there is some possibility that you may be subject to risks that have not yet been identified.

BENEFITS: There are no direct benefits for participating in this study. An indirect benefit to you for participating in this study is the receipt of a health education intervention. This computerized intervention targets behavior change that could potentially help improve your health (or prevent/reduce risky behaviors).

#### **COSTS AND PAYMENTS**

The researchers want your decision about participating in this study to be absolutely voluntary. Yet they recognize that your participation may pose some inconvenience and requires your time. In order to compensate your time you will receive 2 research credits for this initial appointment. You may also be eligible for follow-up assessments online for which you would be paid \$10 (for 1 and 3 months assessments). Those who complete all follow-up assessments will receive a bonus of an additional \$20. Equivalent research credits may be obtained in other ways. Students do not have to participate in this study, or any Psychology Department study, in order to obtain research credit.

If the researchers find new information during this study that would reasonably change your decision about participating, then they will give it to you.

# CONFIDENTIALITY

All information obtained about you in this study is strictly confidential. The results of this study may be used in reports, presentations and publications, but the researcher will not identify you. After data have finished being collected and analyzed, the files tying your name to your responses will be destroyed.

To help us protect your privacy, we have obtained a Certificate of Confidentiality from the National Institutes of Health. The researchers can use this Certificate to legally refuse to disclose information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if there is a court subpoena. The researchers will use the Certificate to resist any demands for information that would identify you, except as explained below.

The Certificate cannot be used to resist a demand for information from personnel of the United States federal or state government agency sponsoring the project, in this case, the National Institutes of Health, and that will be used for auditing or program evaluation of agency funded projects. You should understand that a Certificate of Confidentiality does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If an insurer, medical care provider, or other person obtains your written consent to receive research information, then the researchers will not use the Certificate to withhold that information.

# **WITHDRAWAL PRIVILEGE**

It is OK for you to say NO. Even if you say YES now, you are free to say NO later, and walk away or withdraw from the study -- at any time. Your decision will not affect your relationship with Old Dominion University, or otherwise cause a loss of benefits to which you might otherwise be entitled. The researchers reserve the right to withdraw your participation in this study, at any time, if they observe potential problems with your continued participation.

#### **COMPENSATION FOR ILLNESS AND INJURY**

If you say YES, then your consent in this document does not waive any of your legal rights. However, in the event of harm arising from this study, neither Old Dominion University nor the researchers are able to give you any money, insurance coverage, free medical care, or any other compensation for such injury. In the event that you suffer injury as a result of participation in this research project, you may contact Dr. Abby Braitman at <a href="mailto:abraitma@odu.edu">abraitma@odu.edu</a> or Dr. Michelle Kelley at <a href="mailto:mkelley@odu.edu">mkelley@odu.edu</a> or Dr. Tancy Vandecar-Burdin, the current IRB chair at 757-683-3802 at Old Dominion University, or the ODU Office of Research, at 757-683-3460, who will be glad to review the matter with you.

## **VOLUNTARY CONSENT**

By signing this form, you are saying several things. You are saying that you have read this form or have had it read to you, that you are satisfied that you understand this form, the research study, and its risks and benefits. The researchers should have answered any questions you may have had about the research. If you have any questions later on, then the researchers should be able to answer them:

Abby L. Braitman, Ph.D., abraitma@odu.edu; Michelle L. Kelley, Ph.D., mkelley@odu.edu

If at any time you feel pressured to participate, or if you have any questions about your rights or this form, then you should call Dr. Tancy Vandecar-Burdin, the current IRB chair, at 757-683-3802, or the Old Dominion University Office of Research, at 757-683-3460.

And importantly, by signing below, you are telling the researcher YES, that you agree to participate in this study. The researcher should give you a copy of this form for your records.

#### INVESTIGATOR'S STATEMENT

Subject's Printed Name & Signature

I certify that I have explained to this subject the nature and purpose of this research, including benefits, risks, costs, and any experimental procedures. I have described the rights and protections afforded to human subjects and have done nothing to pressure, coerce, or falsely entice this subject into participating. I am aware of my obligations under state and federal laws, and promise compliance. I have answered the subject's questions and have encouraged him/her to ask additional guestions at any time during the course of this study. I witnessed the above signature(s) on this consent form.

| Investigator's Printed Name & Signature | Date |
|-----------------------------------------|------|